CLINICAL TRIAL: NCT02814292
Title: A Cost-Effective Handheld Breast Scanner for Use in Low Resource Environments: A Validation Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: UE LifeSciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 819121
Record Dates: First submitted 2016-06-14; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Validation of the PEFS to detect breast tumors will be performed by means of a prospective trial. Subjects will participate for 1 clinic visit. Readings from the PEFS will be studied for reproducibility and predictive ability. Data analysis will be iterative, moving on with each modification of the device until the final prototype is created.

DETAILED DESCRIPTION:
Phase 2A of this study is directed primarily at prototype development, creating, testing, and modifying a 4x4 finger array device with a small footprint that is battery powered and reliable. The testing in this phase is aimed at proving that modifications did not degrade the screening sensitivity of the original lab prototype.

Target enrollment is up to 100 patients to verify that the investigators have reproducible values in the same patient. Each breast will be evaluated and compared against each other whether it is considered normal or abnormal tissue. Data from patients both normal and abnormal regions will be compared and used to determine predictive value and accuracy in this prototype. The patient population will be women and men 18 years of age or older with symptomatic breast lump either by palpation or imaging.

Symptomatic individuals scheduled to undergo diagnostic exam will be recruited from all patients presenting for breast evaluations at Dr. Brooks clinical practices who meet all the inclusion and exclusion criteria. Consent will be obtained prior to any study related activities. The PEFS evaluation will be performed by a trained individual. Subjects will be scanned in supine position without breast immobilization - similar to ultrasound testing. The PEFS data is recorded and processed by an automated software algorithm and the results are displayed topographically on a breast-map with red areas showing positive findings and black areas showing negative findings. Quantitative data will be documented and analyzed for accuracy metrics. Results will not be given to subjects nor recorded in their medical records. Because this study is not a clinical utility study, results will have no effect on clinical care decisions. The PEFS evaluation may add between 10 and 30 minutes to the clinic visit. No imaging or pathology tests are being done for research purposes.

ELIGIBILITY:
Inclusion Criteria:

18 years or older

* women or men with symptomatic breast lump by palpation or imaging

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age and older Women and men with symptomatic breast lump either by palpation or imaging
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Estimate the sensitivity of the iBE device examinations using imaging results | through study completion an average of 12 months
Estimate the specificity of the iBE device using imaging results | through study completion an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Broach RB, Geha R, Englander BS, DeLaCruz L, Thrash H, Brooks AD. A cost-effective handheld breast scanner for use in low-resource environments: a validation study. World J Surg Oncol. 2016 Oct 28;14(1):277. doi: 10.1186/s12957-016-1022-2. PMID 27793162